CLINICAL TRIAL: NCT03800953
Title: Chemotherapy/Avelumab Plus Radiotherapy to Primary Esophageal Tumor for Newly Diagnosed Metastatic Esophageal Squamous Cell Carcinoma: The Ave-CRT Study
Brief Title: The Ave-CRT Study for Newly Diagnosed Metastatic Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201809084MIPC
Record Dates: First submitted 2019-01-08; First posted 2019-01-11 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2020-11

CONDITIONS: Esophageal Tumor; Metastatic Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avelumab (Bavencio) (Experimental): This is a single arm, and open label study. All the subjects recruited will receive Avelumab.
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — The study treatment comprises two phases, the concurrent immune-chemoradiotherapy (Ave-PF-CRT) phase and the immune-chemotherapy (Ave-PF) phase. All the subjects will receive Avelumab at both phases.
  Other Names: Bavencio

SUMMARY:
This is a single institutional, single arm, open labeled phase II study to assess the overall radiographic response of adding Avelumab to chemotherapy and palliative radiotherapy in patients with metastatic advanced esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
Avelumab belongs to the group of immune checkpoint blockade cancer therapies. Avelumab binds to the programmed death-ligand 1 (PD-L1) and therefore inhibits binding to its receptor programmed cell death 1 (PD-1). In the case of avelumab, the formation of PD-1/PDL1 ligand pairs is blocked and CD8+ T cell immune response should be increased. This study comprises 2 phases, the concurrent immune-chemoradiotherapy (Ave-PF-CRT) phase and the immune-chemotherapy (Ave-PF) phase. In the immune-chemoradiotherapy phase, patients are treated with PF-CRT and concomitant Avelumab. In the immune-chemotherapy phase, patients are treated with PF plus Avelumab. Overall radiological response, time to progression, overall survival and adverse events will be evaluated. Subjects' health-related quality of life will be assessed as well.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for inclusion, patients must fulfill the following criteria:

  1. Histologically proved squamous cell carcinoma of esophagus
  2. Metastatic disease, which are defined by TNM system of American Joint Committee on Cancer (AJCC) Cancer Staging System (8th edition) in 2017, involving distant lymph node (para-aortic or cervical) metastasis and/or visceral metastasis (lung, liver) documented by radiological examinations
  3. Age ≥ 20 years
  4. ECOG Performance Status 0 or 1
  5. Adequate bone marrow reserves within 2 weeks prior to registration, defined as:a. absolute neutrophil count (ANC) ≥ 1.5×109/L (1,500/μl)b. platelets ≥ 100×109/L (100,000/µl)c. hemoglobin ≥ 9.0 g/dl (may have been transfused)
  6. Adequate liver function reserves within 2 weeks prior to registration, defined as:

     1. hepatic transaminases (AST and ALT) ≤ 2.5 × upper limit of normal (ULN) or ≤ 5 × ULN for subjects with documented metastatic disease to liver
     2. serum total bilirubin ≤ 2.5 × upper limit of normal (ULN)
  7. Adequate renal function within 2 weeks prior to registration: Creatinine ≤1.5 mg/dL
  8. Negative serum or urine pregnancy test for women of childbearing potential
  9. Women of childbearing potential and male participants must practice highly effective contraception throughout the study and for at least 30 days after last avelumab treatment administration if the risk of conception exists
  10. Patients must be able to comply with the study protocol and follow-up schedules and provide study-specific informed consent

Exclusion Criteria:

* Patients fulfill any of the following criteria will be excluded from this trial

  1. Prior radiotherapy to head and neck, chest, or abdomen
  2. Tumor invasion to adjacent structures (T4 lesion)
  3. Adenocarcinoma of esophagus or gastroesophageal junction.
  4. No measurable metastatic target lesion(s) by RECIST criteria
  5. Synchronously or metachronously diagnosed squamous cell carcinoma of aerodigestive way, other than esophageal cancer
  6. Prior invasive malignancy
  7. Prior organ transplantation including allogenic stem-cell transplantation
  8. Current use of immunosuppressive medication, EXCEPT for the following:

     1. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection)
     2. systemic corticosteroids at physiologic doses '≤ 10 mg/day of prednisone or equivalent
     3. steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
  9. Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
  10. Severe, active comorbidities which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and adverse events of the protocol, or limit compliance with study requirements, defined as follows:

      1. Uncontrolled active infection requiring intravenous antibiotics at the time of registration
      2. Transmural myocardial infarction < 6 months prior to registration
      3. Unstable angina or congestive heart failure requiring hospitalization < 6 months prior to registration
      4. Life-threatening uncontrolled clinically significant cardiac arrhythmias
      5. Cerebral vascular accident/stroke (< 6 months prior to enrollment)
      6. Congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
      7. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
      8. Chronic obstructive pulmonary disease exacerbation or other respiratory illness including pulmonary fibrosis requiring hospitalization or precluding study therapy at the time of registration
      9. Uncontrolled psychiatric disorder including recent (within the past year) or active suicidal ideation or behavior
      10. Laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results
      11. Immune colitis, inflammatory bowel disease, immune pneumonitis
  11. Known history of testing positive for HIV or known acquired immunodeficiency syndrome."
  12. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)
  13. Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines
  14. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3)"
  15. Women of childbearing potential and male participants who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the radiation treatment involved in this study may be significantly teratogenic

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
overall radiographic response | 6 months
  overall radiographic response at six-month will be determined by iRECIST

SECONDARY OUTCOMES:
Best radiographic response | up to 2 years
  The best radiographic response of in-field irradiated and out-field non-irradiated (abscopal effect) target lesions will be determined by iRECIST.
Progression-free survival | up to 2 years
  Kaplan-Meier survival estimator will be used to determine the median time to progression for study population (along with 95% confidence interval). The log-rank test will be performed to evaluate the equality of survivor functions across stage, and other covariates of interest on progression-free survival.
Overall survival | up to 2 years
  Kaplan-Meier survival estimator will be used to determine the median time to death for study population (along with 95% confidence interval). The log-rank test will be performed to evaluate the equality of survivor functions across stage, age, and other covariates of interest on overall survival.
Frequency of adverse events | up to 2 years
  The tabulations will count the number of subjects reporting individual adverse events. Adverse events are collected/assessed during treatment period (every week in the Ave-PF-CRT phase [one cycle, 4 weeks], the first and third week of each cycle in the Ave-PF phase [5 cycles, each cycle is 4 weeks]), every 3 months during evaluation, and in 2 years.
Heath-related quality of life | up to 2 years
  The self-reported health-related quality of life specific to esophageal cancer is a 44-item functioning scale captured using the Functional Assessment Of Cancer Therapy-Esophageal (FACT-E) Traditional Chinese version. Each question uses a 5-point Likert scale ranging from 0 to 4, and higher scores indicate better quality of life (0-176 for FACT-E total score). The FACT-E is assessed before treating is given, in the third week of Ave-PF-CRT phase (one cycle, 4 weeks), in the first week of every cycle (4 weeks) during the Ave-PF phase (5 cycles), and in the 2 years.
  Changes in total score of FACT-E from baseline to each assessment point will be calculated.
New metastasis-free survival | up to 2 years
  Kaplan-Meier survival estimator will be used to determine the median time to development of new metastasis for study population (along with 95% confidence interval). The log-rank test will be performed to evaluate the equality of survivor functions across stage, and other covariates of interest on new metastasis-free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsien Cheng, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taiwan, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided